CLINICAL TRIAL: NCT02175940
Title: Effect of Intravitreal Ranibizumab Injection on Aqueous Humor Concentrations of Vascular Endothelial Growth Factor and Pigment Epithelium-derived Factor in Patients With Myopic Choroidal Neovascularization.
Brief Title: VEGF and PEDF in Patients With Myopic Choroidal Neovascularization
Status: Completed | Type: Observational
Sponsor: Università degli Studi di Brescia (Other)
Collaborators: Ciro Costagliola (Unknown); Francesco Semeraro (Unknown); Roberto dell'Omo (Unknown); Mario R Romano (Unknown); Fabiana Aceto (Unknown); Rodolfo Mastropasqua (Unknown); Antonio Porcellini (Unknown)
Responsible Party: Principal Investigator, Andrea Russo, MD, PhD Researcher, Università degli Studi di Brescia
Other Study IDs: VEGF001
Record Dates: First submitted 2014-06-24; First posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Myopic Choroidal Neovascularization; VEGF Aqueous Level; PEDF Aqueous Level

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Myopic Choroidal Neovascularization patients
- Control patients undergoing cataract surgery

SUMMARY:
This was a prospective, case-control study investigating aqueous levels of VEGF and PEDF in eyes with mCNV treated with IVB.

ELIGIBILITY:
Inclusion Criteria:

* pathologic myopia, defined as spherical equivalent >6 diopters and axial length >26 mm
* posterior pole myopic retinal changes (posterior staphyloma, chorioretinal atrophy, papillary crescent);
* fluorescein angiography, indocyanine green angiography and optical coherence tomography detection of the subfoveal or juxtafoveal choroidal neovascularization
* clear ocular media;

Exclusion Criteria:

* previous treatment for choroidal neovascularization, including the previous intravitreal drug injection or PDT
* presence of other maculopathy as diabetic retinopathy or retinal vascular occlusion
* history of recent myocardial infarction or other thromboembolic events
* ongoing uncontrolled hypertension or glaucoma
* refractive media opacities
* previous eye surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with myopic Choroidal Neovascularization treated with intravitreal ranibizumab at the Medical Retina Department, University of Molise, Campobasso, Italy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
vascular endothelial growth factor (VEGF) aqueous levels | 2 months
  VEGF aqueous levels before and after intravitreal ranibizumab
pigment epithelium-derived factor (PEDF) aqueous levels | 2 months
  PEDF aqueous levels before and after intravitreal ranibizumab

SECONDARY OUTCOMES:
best-corrected visual acuity | 2 months
central retinal thickness | 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Retina Department, University of Molise, Cambpobasso, CB, Italy

REFERENCES:
- [Derived] Costagliola C, Semeraro F, dell'Omo R, Romano MR, Russo A, Aceto F, Mastropasqua R, Porcellini A. Effect of intravitreal ranibizumab injections on aqueous humour concentrations of vascular endothelial growth factor and pigment epithelium-derived factor in patients with myopic choroidal neovascularisation. Br J Ophthalmol. 2015 Jul;99(7):1004-8. doi: 10.1136/bjophthalmol-2014-306465. Epub 2015 Mar 13. PMID 25770144